CLINICAL TRIAL: NCT01170104
Title: Phase II Trial of TACE With Sorafenib in Patients With Locally Advanced Hepatocellular Carcinoma
Brief Title: Trial of Transcatheter Arterial Chemoembolization (TACE) With Sorafenib for Locally Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University (Other)
Collaborators: Gyeongsang National University Hospital (Other)
Responsible Party: Joung-Soon Jang/Professor, Chung-Ang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUHHO 2009-1
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sorafenib; TACE; locally, advanced Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sorafenib — Sorafenib (NEXAVAR, Bayer) will be administered after TACE continuous dosing from day 1 until progression or up to 6 cycles of TACE as an oral 400mg twice-daily without food (at least 1 hour before or 2 hours after eating).
Procedure: TACE (Transcatheter arterial chemoembolization) — Sorafenib (NEXAVAR, Bayer) will be administered after TACE continuous dosing from day 1 until progression or up to 6 cycles of TACE as an oral 400mg twice-daily without food (at least 1 hour before or 2 hours after eating).

SUMMARY:
To evaluate the time to progression of the combination therapy of Transcatheter Arterial Chemoembolization (TACE) and sorafenib in patients with previously untreated advanced or metastatic hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable Hepatocellular carcinoma with local liver lesion treatable with TACE
2. Age > 18 years.
3. ECOG Performance Status of 0 or 1.
4. Child-Pugh class A (class B could be included when Childs score is 7).
5. Life expectancy of at least 12 weeks.
6. Subjects with at least one measurable lesion.
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   * Hemoglobin > 9.0 g/dl
   * Absolute neutrophil count (ANC) >1,500/mm3
   * Platelet count > 75,000/μl
   * Total bilirubin < 1.5 times the upper limit of normal
   * ALT and AST < 2.5 x upper limit of normal (UNL)
   * Alkaline phosphatase < 5 x ULN
   * PT-INR/PTT < 1.5 x upper limit of normal
   * Serum creatinine < 1.5 x ULN
8. Signed and dated informed consent before the start of specific protocol procedures

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy( beta blockers or digoxin are permitted) or uncontrolled hypertension.
2. History of HIV infection.
3. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
4. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
5. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
6. History of organ allograft The organ allograft may be allowed as protocol specific.
7. Patients with evidence or history of uncontrolled bleeding diathesis
8. Patients undergoing renal dialysis
9. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
10. Excluded therapies and medications, previous and concomitant:

    * Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry
    * Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed). Major surgery within 4 weeks of start of study
    * Investigational drug therapy outside of this trial during or within 4 weeks of study entry
    * Prior exposure to the study drug.
    * Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial (and men for at least 3 months after last administration of study medication).
    * Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
    * Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
    * Patients unable to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 2 year
  Assessments including image and laboratory studies will take place within 7days of the every TACE cycle

SECONDARY OUTCOMES:
To evaluate the toxicity profiles | 2 year
  Clinically assessed every TACE cycle

CONTACTS AND LOCATIONS:
Overall Officials: Joung-Soon Jang, M.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hospital, Dongjak, Seoul, South Korea